CLINICAL TRIAL: NCT02788409
Title: Incidence of Second Primary Malignancies in Patients With Castration-Resistant Prostate Cancer: An Observational Retrospective Cohort Study in the US
Brief Title: Incidence of Second Primary Malignancies in Castration-Resistant Prostate Cancer: An Observational Retrospective Cohort Study in the US
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: 18673
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medicare CRPC: Men in the US older than 65 years old having CRPC
  Interventions: Other: Not applicable for study

INTERVENTIONS:
Other: Not applicable for study — Provide external perspective on background second primary cancer incidence rates for REASSURE study.

SUMMARY:
This study is conducted to estimate population-based incidence rates of second primary malignancies among patients with CRPC similar to those treated with Xofigo. These rates will provide context for second primary malignancy incidence rates from the REASSURE study.

Furthermore this study aims to provide further information about the documentation of bone metastases in Medicare data and the extent of use of only oral androgen deprivation drugs among patients with Medicare Part D coverage, as well as to estimate overall survival of the study population.

DETAILED DESCRIPTION:
Xofigo (radium-223 dichloride) is an alpha-emitting pharmaceutical, which was approved for the treatment of patients with castration-resistant prostate cancer (CRPC), symptomatic bone metastases, and no known visceral metastatic disease. The long-term safety profile of Xofigo is evaluated in the prospective REASSURE study, which estimates the incidence rates of second primary malignancies in patients with CRPC receiving Xofigo.

To provide context on that, this retrospective study is conducted to estimate background rates of second primary malignancies among patients with CRPC similar to those who are treated with Xofigo.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in both Medicare Parts A and B for at least 1 year before the cohort entry date (minimum lookback period for comorbidities and treatments)
* Primary site code of prostate cancer (International Classification of Diseases for Oncology, Third Edition [ICD-O-3] topography code C61.9) in SEER data
* Surgical castration or androgen deprivation therapy after prostate cancer diagnosis; androgen deprivation therapy will be indicated by the use of any of the following drugs: abarelix, bicalutamide, buserelin, cyproterone, degarelix, diethylstilbestrol, estramustine, flutamide, gonadorelin, goserelin, histrelin, leuprolide, medroxyprogesterone, megestrol, nafarelin, nilutamide, polyestradiol, triptorelin
* Evidence that prostate cancer was resistant to surgical castration or androgen deprivation therapy ("castration-resistant prostate cancer"), as indicated by starting one of the following second-line systemic therapies (cohort entry date): abiraterone, cabazitaxel, docetaxel, enzalutamide, mitoxantrone, or sipuleucel-T
* Cohort entry date 01 January 2006 or later
* Age 65 years or older in the US on the cohort entry date

Exclusion Criteria:

* Enrollment in an HMO (Health Maintenance Organization) in the year before the cohort entry date
* Diagnosis of any cancer other than prostate cancer or nonmelanoma skin cancer on or before the cohort entry date
* Any diagnostic code for metastases other than bone metastases or lymph node metastases on or before the cohort entry date
* Any claim for treatment with Xofigo on or before the cohort entry date.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The cohort will include men who are enrolled in both Medicare Parts A and B for at least 1 year before the cohort entry date, have a primary site code of prostate cancer in SEER data, have surgical castration or androgen deprivation therapy after prostate cancer diagnosis, have evidence that prostate cancer was resistant to the castration as indicated by starting a second-line systemic therapy, and have an cohort entry date of 01 January 2006 or later on which they are aged 65 years or older. All eligible subjects will be selected; there will be no sampling. (The probability of selecting each eligible patient is equal to 1)
Sampling Method: Probability Sample
Enrollment: 2234 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence rate of second primary malignancy | Retrospective analysis between 1-Jan-2000 and 31-Dec-2013
Incidence rates of skeletal-related events | Retrospective analysis between 1-Jan-2000 and 31-Dec-2013

SECONDARY OUTCOMES:
Proportion with a history of bone metastasis at cohort entry | Retrospective analysis between 1-Jan-2000 and 31-Dec-2013
Proportion who met the definition of castration based solely on Part D data | Retrospective analysis between 1-Jan-2000 and 31-Dec-2013
Overall survival | Retrospective analysis between 1-Jan-2000 and 31-Dec-2013

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Waltham, Massachusetts, United States